CLINICAL TRIAL: NCT02231073
Title: Peripheral and Central Postural Disorders in the Elderly
Brief Title: Exercise, Brain Imaging, Cognition, and Gait in Parkinsonism
Acronym: EEforPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Fay B. Horak, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 4131; 2R01AG006457 (NIH)
Record Dates: First submitted 2014-08-18; First posted 2014-09-04 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Parkinson's Disease
Keywords: Freezing of gait; Idiopathic Parkinson's disease; Exercise; parkinsonism
MeSH Terms: conditions — Parkinson Disease; Motor Activity; Parkinsonian Disorders | interventions — Exercise; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise: Agility Boot Camp-Cognitive (Experimental): Subjects will participate in an 80-minute, group (6 per group) exercise session led by a certified exercise trainer knowledgeable in the Agility Boot Camp-Cognitive (ABC-C) program for 3x/week for 6 weeks. The exercise protocol is an adaptation of our Agility Boot Camp (ABC) exercise program for PD. The exercises are designed as a circuit to challenge movement-skills known to be impaired in PD. Stations will include: Gait training, PWR Moves ©, Agility course, Lunges, Boxing and Tai Chi. Each activity was chosen for its inherent focus on multi-directional movements, dynamic postural transitions, axial mobility, big movements and whole body motor sequencing. Each station (10-20 minutes) has 3 possible progression levels, based on: (1) divided attention with secondary cognitive tasks, (2) response inhibition, (3) limiting external sensory cues, and (4) increasing speed and resistance.
  Interventions: Behavioral: Exercise and Education for Parkinson's Disease
- Education: Living with Parkinson's disease (Active Comparator): The Education arm is a chronic disease education program to teach patients how to live better with their chronic condition. It was developed by our research team to be specific for people with Parkinson's disease. It will include content and discussion of topics such as sleep, nutrition, and medication management. Classes will consist of a group of subjects (up to 6) meeting with the trainer for 90-minute session, once a week for six weeks. In order to match dose of the education intervention with the exercise intervention, participants will be provided relaxation tapes to be used at home 5 times per week for 30 minutes for an overall education dose of 240 minutes; similar to the exercise dose.
  Interventions: Behavioral: Exercise and Education for Parkinson's Disease

INTERVENTIONS:
Behavioral: Exercise and Education for Parkinson's Disease — Exercise and Education for Parkinson's Disease for 6 week cross-over intervention.

SUMMARY:
There is emerging research detailing the relationship between balance/gait/falls and cognition. Imaging studies also suggest a link between structural and functional changes in the frontal lobe (a region commonly associated with cognitive function) and mobility. People with Parkinson's disease have important changes in cognitive function that may impact rehabilitation efficacy. Our underlying hypothesis is that cognitive function and frontal lobe connections with the basal ganglia and brainstem posture/locomotor centers are responsible for postural deficits in people with Parkinson's disease and play a role in rehabilitation efficacy. The purpose of this study is to 1) determine if people with Parkinson's disease can improve mobility and/or cognition after partaking in a cognitively challenging mobility exercise program and 2) determine if cognition and brain circuitry deficits predict responsiveness to exercise rehabilitation.

Design: This study is a randomized cross-over controlled intervention to take place at a University Balance Disorders Laboratory. The study participants will be people with Parkinson's disease who meet inclusion criteria for the study. The intervention will be 6 weeks of group exercise (case) and 6 weeks of group education (control). The exercise is a cognitively challenging program based on the Agility Boot Camp for people with PD. The education program is a 6-week program to teach people how to better live with a chronic disease. The primary outcome measure is the MiniBESTest and the secondary outcomes are measures of mobility, cognition and neural imaging.

Discussion: The results from this study will further our understanding of the relationship between cognition and mobility with a focus on brain circuitry as it relates to rehabilitation potential.

ELIGIBILITY:
Inclusion criteria:

Aged 50-90 years old. No musculoskeletal or peripheral or central nervous system disorders (other than idiopathic Parkinson disease (iPD) or parkinsonism) that could significantly affect balance or gait .

Capable of following directions. iPD subjects: UK Brain Bank criteria, i.e., bradykinesia and at least one of the following: rest tremor, muscular rigidity, and postural instability not cause by visual, vestibular, cerebellar or proprioceptive dysfunction. Unilateral onset, response to levodopa.

Parkinsonism subjects: Gait characterized by slow short steps, shuffling gait and may be wide-based, with FoG, postural instability.

Exclusion criteria:

Inability to stand or walk for 2 min without an assistive device Recent changes in medication Excessive use of alcohol or recreational drugs, Contraindications to MRI scans (eg, claustrophobia, metal in body) Intervention subjects will be excluded if: 1) participating in a vigorous exercise program more than 2 x/week, 2) A medical condition that contraindicates exercise participation.

Parkinsonism subjects: iPD and Parkinson plus syndromes such as Progressive Supranuclear Palsy, Multiple System Atrophy, Corticobasal Syndrome, or Cerebellar Ataxia.

Idiopathic PD subjects: Same as above and deep brain stimulation electrodes. Significant tremor that would interfere withMRI scan.

Control subjects: Will be matched for age and gender to iPD and parkinsonism groups.

-

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Change in Mini-BESTest score | Three timepoints; baseline, 6 weeks (after Arm 1), 12 weeks (after Arm 2)
  The Mini-BESTest assesses dynamic balance via a 14-item test that measures multiple domains of balance including anticipatory postural adjustments, reactive postural control, sensory orientation, dynamic gait.

SECONDARY OUTCOMES:
Change in MDS-UPDRS score | Three timepoints; baseline, 6 weeks (after Arm 1), 12 weeks (after Arm 2)
  The Unified Parkinson's Disease Rating Scale Motor Subscale III is a 10-minute assessment of motor signs related to severity of PD. If the investigators have trouble recruiting subjects of similar severity in the 2 groups, they will use the Postural Instability and Gait Disability(PIGD) Subscore (Items 27-30) as a covariate in data analysis.
Change in New Freezing of Gait questionnaire (NFOGQ) score | Three timepoints; baseline, 6 weeks (after Arm 1), 12 weeks (after Arm 2)
  The New FoG of Gait Questionnaire will be used to identify 'freezers' (score >3). NFOGQ is a self-report measure that begins with the presentation of a short (30-s) video to illustrate FoG during walking turning and starting gait and then follows with questions related to frequency and duration of each type of FoG episode.
Change in PDQ-39 score | Three timepoints; baseline, 6 weeks (after Arm 1), 12 weeks (after Arm 2)
  the Parkinson's Disease Quality of Life questionnaire with 39 questions reflecting 8 domains of quality of life (Mobility, ADL's, Emotional well-being, Stigma, Social support, Cognition, Communication, and Bodily discomfort). Each item scores from 0 (never) to 4 (always). Subscale scores and a summary index representing the global health-related quality of life will be calculated, with higher scores representing worse quality of life. Convergent validity is very good and discriminative validity for PD severity levels has been established. The PDQ will reflect limitations to participation in community mobility.
Change in Activities of Balance Confidence (ABC) questionnaire score | Three timepoints; baseline, 6 weeks (after Arm 1), 12 weeks (after Arm 2)
  Activities of Balance Confidence (ABC) questionnaire consists of 16 questions about how balance confidence limits participating in the community such as riding an escalator, walking in a parking lot and replacing a light. Subjects indicate their confidence from 0% to 100% they have in their balance when they imagine doing these tasks. A score of 80% indicates an average level of physical functioning for older adults.
Change in instrumented gait and balance measures | Three timepoints; baseline, 6 weeks (after Arm 1), 12 weeks (after Arm 2)
  Balance: Postural sway during quiet stance with and without a cognitive task. Gait: Spatial and temporal gait metrics will be collected during walking, while wearing the Opal inertial sensors, with and without a cognitive task.
  Turning: Smoothness of turning measure during 1 min turning in place (360 degree) and turns during 2 min walk, with and without a cognitive task.
Neural Imaging | Baseline
  DTI: High angular resolution diffusion imaging to assess white matter microstructure. Structural connectivity of the locomotor network will be assessed using probabilistic tractography.
  rsfcMRI: An indirect assessment of communication between spatially disparate neural regions. Analysis is restricted to neural regions comprising the locomotor network including the supplementary motor area, subthalamic nuclei, mesencephalic locomotor regions (pedunculopontine and cuneiform nuclei), and the midline cerebellar locomotor region
Change in Cognitive measures | Three timepoints; baseline, 6 weeks (after Arm 1), 12 weeks (after Arm 2)
  A battery of tests to measure different cognitive domains: inhibition (stroop, flankers, go/nogo, stop signal), shifting (set-shifting, trail making), updating (dot counting task), visual-spatial (judgement of line orientation), general cognition (SCOPA-COG), and other (social norms questionnaire, social behavior rating scale, simple reaction time test).

CONTACTS AND LOCATIONS:
Overall Officials: Fay B Horak, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] King LA, Peterson DS, Mancini M, Carlson-Kuhta P, Fling BW, Smulders K, Nutt JG, Dale M, Carter J, Winters-Stone KM, Horak FB. Do cognitive measures and brain circuitry predict outcomes of exercise in Parkinson Disease: a randomized clinical trial. BMC Neurol. 2015 Oct 24;15:218. doi: 10.1186/s12883-015-0474-2. PMID 26499867